CLINICAL TRIAL: NCT00485368
Title: The Effect of an Angiotensin Converting Enzyme Inhibitor on Aortic Wall Properties in Patients With Marfan Syndrome.
Brief Title: Angiotensin Converting Enzyme Inhibitors in Marfan Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Baker Heart Research Institute (Other); The Alfred (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3/03
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Marfan Syndrome
Keywords: marfan syndrome; aortic root diameter
MeSH Terms: conditions — Marfan Syndrome | interventions — Perindopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Coversyl (perindopril)

SUMMARY:
The purpose of this research is to assess the effects of a drug called perindopril on the aorta in people known to have Marfan Syndrome. The aorta is the major artery of the body that comes out of the heart and supplies blood to the body. We know that in people with Marfan Syndrome, the aorta is stiff and this stiffness results in its enlargement over many years. This enlargement of the aorta can be very serious. We know from treatment of other heart conditions that drugs of the same type as perindopril reduce stiffness of the arteries. This type of drug has never been tried in people with Marfan Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* Diagnosis of Marfan Syndrome, on the basis of the Ghent Criteria

Exclusion Criteria:

* Age <18, >40
* Women of child-bearing potential not on adequate contraception
* Serum creatinine of >0.11
* A history of intolerance to ACEI
* Patients on angiotensin receptor blockers
* Blood pressure >140/90mmHg
* History of previous aortic surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2004-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
aortic root diameter | 24 weeks

SECONDARY OUTCOMES:
arterial stiffness | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn A Kingwell, PhD, Principal Investigator — Baker Heart Research Institute

REFERENCES:
- [Derived] Ahimastos AA, Aggarwal A, D'Orsa KM, Formosa MF, White AJ, Savarirayan R, Dart AM, Kingwell BA. Effect of perindopril on large artery stiffness and aortic root diameter in patients with Marfan syndrome: a randomized controlled trial. JAMA. 2007 Oct 3;298(13):1539-47. doi: 10.1001/jama.298.13.1539. PMID 17911499 (Retraction: PMID 26594834 JAMA. 2015 Dec 22-29;314(24):2692-3)